CLINICAL TRIAL: NCT04320329
Title: Natural History of Morquio B and Late-Onset GM1 Gangliosidosis
Brief Title: Natural History of Morquio B and Late-Onset of GM1 Gangliosidosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other); Medical University of Graz (Other)
Responsible Party: Principal Investigator, Sylvia Stockler, MD, PhD, MBA, FRCPC, University of British Columbia
Other Study IDs: H18-00155
Record Dates: First submitted 2020-03-17; First posted 2020-03-25 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Morquio B Disease; GM1 Gangliosidosis Type III
MeSH Terms: conditions — Mucopolysaccharidosis IV; Gangliosidosis, GM1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Urine Dried Blood Spot sample Fibroblasts frozen live cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mucopolysaccharidosis type IVB (Morquio-B disease, MBD) is an autosomal-recessive lysosomal disease caused by mutations in a gene called GLB1. Clinically, Morquio B presents with progressive skeletal deformities involving mostly long bones and spine. While the information on GLB1 mutations associated with MBD is limited, there is a significant overlap in clinical presentation between Morquio B and late-onset GM1 gangliosidosis with both conditions being caused by mutations in the same GLB1 gene. In this study, the investigators plan to collect retrospective data from patients' medical charts, as well as, information from the prospective follow up clinic visits. There will be two study visits with the interval of one year. The study procedures will include a detailed physical exam, bone scans, heart and lung function, physical endurance tests, hearing test, laboratory tests and quality of life surveys.

The purpose of this study is to collect data on the natural history of Morquio B and to create a biobank of laboratory samples (blood, urine and skin cells) for future research. This information will improve the understanding of the natural progression of Morquio B disease.

DETAILED DESCRIPTION:
The primary objective of this study is to establish the natural history of Morquio B (Mucopolysaccharidosis type IVB, MBD) disease through the collection and analysis of retrospective and prospective data on patients diagnosed with Morquio B. Because of significant overlap in clinical presentation, patients with late-onset GM1 will also be included.

Upon consent, data from clinical, laboratory, functional and quality of life studies, and data from review of medical records will be collected and analyzed descriptively. In addition, the samples of blood, urine and fibroblasts will be collected and stored at BC Children Hospital Research Institute Biobank for future research. The prospective follow up will include two clinic visits, one year apart. The following data will be collected during the prospective observational part of the study (as per study protocol) and retrospective part (whether such data are available from the medical chart):

* Medical history: Morquio B / Late-onset GM1 gangliosidosis diagnosis, presentation, treatments and symptom progression
* Physical exam, including neurological and ophthalmological assessments
* Standard Grip Strength Evaluation
* Range of motion
* Six-minute walk test (6MWT)
* 3-Minute Stair Climb Test
* Gait and Motion assessment
* Pulmonary function testing
* Hearing test
* Echocardiography
* EKG
* X-ray (lumbar spine, upper & lower limbs, hip)
* DXA scan
* Brain MRI
* Laboratory tests (GAGs assay and pro-inflammatory cytokine panel)
* Blood, urine and fibroblast samples for biobanking
* Genetic test (if not done per standard of care)

Additional assessments and evaluations:

• Patient-reported outcomes: quality of life SF-36, MPS HAQ and the interview on personally meaningful outcomes

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of beta-galactosidase deficiency via demonstration of deficient enzyme activity and/or demonstration of homozygous/compound heterozygous pathogenic GLB1 variants;
* Patients diagnosed with beta-galactosidase deficiency and who present with "MPSIVB skeletal phenotype" with or without primary CNS involvement;
* Patient / parent or legal guardian is able to read, understand, and sign the informed consent.

Exclusion Criteria:

* Previous Hematopoietic Stem Cell Transplant procedure (HSCT);
* Concurrent disease or condition that would interfere with participation in the study and/or travel to the site (for the prospective follow up);
* Previous or current casual treatments that might affect the natural course of the disease;
* Patient's (guardian's) not understanding and/or not agreeing to the informed consent form;
* GM1-gangliosidosis patients who present without "MPSIVB skeletal phenotype"

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age, any gender with no previous HSCT procedure, with a confirmed diagnosis of beta-galactosidase deficiency and who clinically present with skeletal dysostosis with or without CNS involvement.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Physical Development | Through study completion, an average of 1 year
  Height
Physical Development | Through study completion, an average of 1 year
  Weight
Physical Development | Through study completion, an average of 1 year
  Growth rate
Physical Endurance | 1 year
  6MWT
Physical Endurance | 1 year
  3MSCT
Physical Endurance | 1 year
  Standard Grip Strength evaluation
Range of Motion Scale | Through study completion, an average of 1 year
  Assessments: shoulder, elbow, wrist, hip, knee, ankle
Skeletal involvement | Through study completion, an average of 1 year
  X-ray studies, pQCT (where available), DXA of lateral distal femur, x-ray and/or MRI of cervical spine to assess spinal stenosis and spinal cord compression; X-ray of cervical spine to assess odontoid hypoplasia and atlantoaxial instability
CNS involvement | Through study completion, an average of 1 year
  Neurological assessments, Brain MRI
Surrogate biomarkers | Baseline and 1 year
  Glycosaminoglycans (GAGs): keratan sulfate, heparan sulfate, dermatan sulfate, chondroitin-6-sulfate
Surrogate biomarkers | Baseline and 1 year
  Comprehensive pro-inflammatory cytokine panel with markers of bone turnover
Health-related Quality of Life (HRQoL) | Baseline and 1 year
  SF-36
Health-related Quality of Life (HRQoL) and Activities of Daily living (ADLs) | Baseline and 1 year
  MPS-HAQ
Personally Meaningful Outcomes | Baseline and 1 year
  PMO Questionnaire

OTHER OUTCOMES:
Biobank of samples for the future research | 1 year
  Blood, urine, DBS, fibroblasts (live frozen cells)

CONTACTS AND LOCATIONS:
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada